CLINICAL TRIAL: NCT00889967
Title: An International, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Once Daily Administration of Two Strengths of Ciprofloxacin for Inhalation Compared With Placebo for Inhalation in the Management of Pseudomonas Aeruginosa in Patients With Non Cystic Fibrosis Bronchiectasis
Brief Title: Safety and Efficacy Study of Ciprofloxacin for Inhalation in Patients With Non-Cystic Fibrosis Bronchiectasis "ORBIT-1"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aradigm Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARD-3100-0901
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2012-08

CONDITIONS: Non-Cystic Fibrosis Bronchiectasis
Keywords: Pseudomonas aeruginosa; antimicrobial; inhalation; ciprofloxacin; Non-Cystic Fibrosis Bronchiectasis
MeSH Terms: conditions — Pseudomonas Infections; Respiratory Aspiration | interventions — Ciprofloxacin; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Ciprofloxacin for Inhalation 100 mg/day by inhalation
  Interventions: Drug: Ciprofloxacin for Inhalation
- 2 (Experimental): Ciprofloxacin for inhalation 150 mg/day by inhalation
  Interventions: Drug: Ciprofloxacin for Inhalation
- Placebo (Placebo Comparator): Placebo by inhalation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin for Inhalation — 100 mg once daily by inhalation for 28 days
  Arms: 1
Drug: Ciprofloxacin for Inhalation — 150 mg once daily by inhalation for 28 days
  Arms: 2
Drug: Placebo — Placebo once daily by inhalation for 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Ciprofloxacin for Inhalation in the treatment of patients with non-cystic fibrosis (CF) bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

1. Are willing and able to provide written informed consent.
2. Are males or females 18 to 80 year of age, inclusive.
3. Have had a confirmed diagnosis of non-CF bronchiectasis per high resolution computed tomography (HRCT) for at least 4 years.
4. Confirmation of infection with P. aeruginosa at screening

Exclusion Criteria:

1. Have a known local or systemic hypersensitivity to fluoroquinolone or quinolone antibiotics.
2. Have an exacerbation during the Screening Phase as defined as requiring treatment with inhaled, oral, or intravenous antibiotics prior to the first dose of study drug.
3. Have a diagnosis of cystic fibrosis..
4. Have had changes in either the treatment regimen or initiation of treatment with any of the following medications within 28 days prior to Visit 1:

   * Azithromycin
   * Hypertonic saline
   * Bronchodilator medications
   * Oral corticosteroid.
5. Have received an investigational drug or device within 28 days prior to Visit 1.
6. Have any serious or active medical or psychiatric illness, which in the opinion of the investigator, would interfere with patients' treatment, assessment, or compliance with the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is defined as the mean change in P. aeruginosa density in sputum (log10) CFU/gram of sputum from Baseline to Day 28. | 28 days

SECONDARY OUTCOMES:
Microbiological efficacy | 28 days
Time to, number of, severity of, and time to resolve exacerbations | 28 days
Changes in spirometry 4. Quality of life (QOL) 5. Safety and tolerability | 28 days
Quality of life (QOL) | 28 days
Safety and tolerability | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bruinenberg, MBChB, MBA, Study Director — Aradigm Corporation
Locations (36):
- United States (14):
  - Phoenix, Arizona
  - Los Angeles, California
  - Sacramento, California
  - Torrance, California
  - Waterbury, Connecticut
  - Brandon, Florida
  - Miami, Florida
  - Council Bluffs, Iowa
  - Summit, New Jersey
  - New York, New York
  - Elizabeth City, North Carolina
  - Toledo, Ohio
  - Philadelphia, Pennsylvania
  - McKinney, Texas
- Canada (6):
  - Calgary, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Montreal, Quebec
  - Saint-Jérôme, Quebec
- Germany (4):
  - Berlin
  - Donaustauf
  - Heidelberg
  - Neuwied
- United Kingdom (12):
  - "Ground Floor, Tower Block, Lisburn Road, Belfast, Britain
  - "1st Floor, Nuffield House, B15 2TH, Birmingham, Britain
  - "Duckworth Lane,, Bradford, Britain
  - "Southmoor Road, M23 9LT, Manchester, Britain
  - Newcastle upon Tyne, Freeman Road, High Heaton
  - London, High Street Lewisham
  - "Bordesley Green East, Birmingham
  - "133 Balornock Road, Glasgow
  - Royal Brompton Hospital, London
  - "Stott Lane, Salford
  - "Newcastle Road, Stoke-on-Trent
  - "Northumbria Healthcare, Tyne and Wear